CLINICAL TRIAL: NCT07219667
Title: Community-Engaged Approach to Supporting South Asians With Type 2 Diabetes at Risk for Depression
Brief Title: South Asians With Type 2 Diabetes at Risk for Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-00438; 1K01DK140613-01A1 (NIH)
Record Dates: First submitted 2025-10-21; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult South Asian patients in the New York City (NYC) region (Experimental): In Aim 3, CHWs will provide culturally and linguistically tailored health education to South Asian participants on the management of T2D and depressive symptoms.
  Interventions: Behavioral: CHW-led T2D Intervention

INTERVENTIONS:
Behavioral: CHW-led T2D Intervention — CHW-led T2D intervention that includes mental health and digital health components.

SUMMARY:
This study will adapt a community health worker (CHW)-led Type 2 diabetes (T2D) intervention to include mental health and digital components using a trauma informed care approach, and test the feasibility and acceptability of this intervention to support South Asians with T2D at risk for depression.

DETAILED DESCRIPTION:
Specific Aim 1: Examine factors associated with distress, poor mental health, and comorbid T2D and depression among South Asians to inform pilot study structure and content.

Specific Aim 2: Adapt CHW-led T2D intervention to include mental health and digital components using a trauma-informed care approach and the ecological validity model.

Specific Aim 3: Evaluate the feasibility and acceptability of a pilot CHW-led intervention to support participants with T2D who are at risk for depression.

ELIGIBILITY:
Inclusion Criteria:

Aim 1 (Qualitative Component):

* South Asian ethnicity based on self-report information
* 18 years of age or older
* Residing in NYC
* Willingness and capacity to provide consent

Aim 3: Pilot Intervention:

* South Asian ethnicity based on patient demographic information
* 18 to 75 years of age
* Appointment for routine non-emergent primary care in the past 12 months
* Diagnosis of Type 2 diabetes
* Patient Health Questionnaire-9 (PHQ-9) score of ≥5 (mild to severe depression)
* Residing in NYC
* Willingness and capacity to provide consent

Exclusion Criteria:

Aim 1 (Qualitative Component):

• Diagnosed cognitive deficits or limited decision-making capacity

Aim 3: Pilot Intervention:

* Pregnant at the time of screening
* Type 1 diabetes or diabetes secondary to other conditions (e.g., steroid-induced, pancreatic insufficiency)
* Malignancy or life-threatening illness with a life expectancy of <5 years
* Inability to perform unsupervised physical activity
* Diagnosed cognitive deficits or limited decision-making capacity
* Currently taking anti-depressant medication or receiving counseling services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c Levels | Baseline, Month 3
  Change in glycated hemoglobin (HbA1c).
Change in Diabetes Distress Scale (DDS) Score | Baseline, Month 3
  The Diabetes Distress Scale (DDS) is a 17-item psychological questionnaire designed to assess the emotional and psychological distress experienced by individuals with diabetes. Each item is rated on a scale of 0 to 6. The total score is calculated by summing up the scores of all 17 items and ranges from 0-102; higher scores indicate greater distress.
Change in Patient Health Questionnaire-9 (PHQ-9) Score | Baseline, Month 3
  The PHQ-9 is a 9-item questionnaire to assess depressive symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27. Higher scores indicate greater severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Naheed Ahmed, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared with researchers who provide a methodologically sound proposals, provided the requesting researcher executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Study data will be deposited into the repository at the time of an associated study publication or end of performance period, whichever comes first. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Study data will be deposited into the repository at the time of an associated study publication or end of performance period, whichever comes first.
Access Criteria: Data are available for 5 years at a third party website (Link to be included).